CLINICAL TRIAL: NCT07255339
Title: The Effect of Music Therapy on Pain and Anxiety in Patients After Coronary Artery Bypass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Tuğba Albayram, Research Assistant Dr, University of Gaziantep
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/17-03
Record Dates: First submitted 2025-11-15; First posted 2025-12-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Music Therapy; Pain; Anxiety; Randomised Controlled Trial; Coronary Artery Bypass Grafting
Keywords: Coronary artery bypass grafting; Music therapy; Pain; Anxiety; Randomized controlled trial
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy group (Active Comparator): Music therapy group
  Interventions: Other: Music therapy group
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Music therapy group — In the study, patients undergoing coronary artery bypass graft surgery will be exposed to music before and during surgery. The Beck Anxiety Inventory and Visual Analog Scale will be administered postoperatively.
  Arms: Music therapy group

SUMMARY:
Coronary artery disease is a frequently occurring, life-threatening disease that has caused high morbidity and mortality, and has resulted in a high rate of death, both in our country and worldwide over the past five years. The most commonly used method for the treatment of coronary artery disease is coronary artery bypass grafting (CABG). This surgery aims to restore blood flow to the myocardium, which has become inadequate due to blockage or stenosis in the coronary arteries that feed the heart, by using an artery graft and to prolong life to a better standard. Surgical procedures such as coronary artery bypass grafting are psychologically, economically, socially, and physically detrimental to patients. Coronary artery bypass grafting, a major surgical procedure, can lead to serious postoperative complications. Some of these include postoperative pain and anxiety. Pain is one of the first complications observed, especially in the early postoperative period. The heart is one of the most important vital organs, and interventions in this regard trigger a fear of death in individuals and, consequently, cause them to experience significant anxiety after the operation. In addition to pharmacological methods, non-pharmacological methods are also used in pain and anxiety management. Music therapy is one of these methods used in the treatment of pain and anxiety. Music has always been a cultural and universal heritage of societies, present from past to present. Music therapy is a specialized field that incorporates the patient's body, mind, and spirit integrity, facilitates treatment using evidence-based practices, and utilizes all aspects of music within a therapeutic relationship to alleviate patient distress. Music therapy has consistently been a part of treatment methods from past to present and has been shown to have positive effects. Depression can affect stress hormones, leading to an increase in heart rate and an imbalance in oxygen demand. Disruption of sleep patterns before surgery can lead to anxiety and pain. Previous studies have shown that music therapy balances the body, mind, and spirit integrity of individuals within the endocrine and nervous systems.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) has remained one of the leading causes of high morbidity and mortality both in our country and worldwide over the past five years. According to global epidemiological data, cardiovascular diseases account for nearly one-third of all deaths, making them a major public health concern. CAD is characterized by atherosclerotic plaque formation and the narrowing of coronary vessels, which results in reduced myocardial oxygenation. As the disease progresses, coronary artery bypass grafting (CABG) becomes one of the most commonly used and effective treatment methods. The primary goal of CABG is to restore myocardial blood flow distal to the stenotic or occluded coronary artery by using arterial or venous grafts, thereby improving cardiac perfusion and enhancing both quality of life and overall survival.

CABG is a major surgical intervention that imposes significant psychological, physiological, social, and economic burdens on patients. In the postoperative period, patients frequently experience severe pain, anxiety, sleep disturbances, stress, depressive symptoms, hemodynamic instability, and reduced quality of life. The intensity of postoperative pain is affected by the invasiveness of the procedure, such as sternotomy, placement of chest tubes, surgical drains, and limited mobility. Moreover, undergoing a surgical procedure involving the heart-a vital organ-often triggers fear of death, a sense of loss of control, uncertainty about recovery, and concerns about postoperative complications, all of which contribute to heightened anxiety levels.

While pharmacological treatments are essential in managing postoperative pain and anxiety, they are often insufficient on their own. For this reason, non-pharmacological interventions are increasingly recommended as complementary approaches during the recovery process. Among these interventions-such as breathing exercises, relaxation techniques, massage therapy, and aromatherapy-music therapy has gained particular attention due to its demonstrated benefits.

Music therapy is a specialized, evidence-based discipline that utilizes the therapeutic elements of music within a structured patient-therapist relationship to support the individual's physical, psychological, and spiritual well-being. By employing components such as rhythm, melody, and harmony, music therapy aims to regulate emotional responses and promote healing. Studies have shown that music has significant effects on the autonomic nervous system; it activates the parasympathetic system, helping to stabilize heart rate, reduce blood pressure, regulate breathing, and decrease levels of stress-related hormones, including cortisol. Consequently, music therapy alleviates both the perception of pain and anxiety.

Furthermore, disruptions in sleep patterns prior to surgery can exacerbate anxiety and pain, while chronic stress and elevated stress hormones may negatively affect heart rate, oxygen demand, and overall cardiopulmonary stability. Previous research has demonstrated that music therapy can help regulate the mind-body-spirit connection within the endocrine and nervous systems, thereby promoting physiological balance and emotional comfort in individuals undergoing major surgical procedures such as CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with no hearing impairment
* Planned for coronary artery bypass graft surgery
* Not diagnosed with a psychiatric disorder and therefore not taking medication
* Volunteer to participate in the study

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients who volunteer to participate and then withdraw from the study at any stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
The effect of music played on anxiety in patients undergoing coronary artery bypass graft surgery | From enrollment to the end of treatment at one years
  "Not at all" indicates no anxiety at all, while "I had a very hard time tolerating it at a serious level" indicates the highest possible anxiety.
The effect of music played on pain in patients undergoing coronary artery bypass graft surgery | From enrollment to the end of treatment at one years
  Zero is equivalent to no pain, and 10 indicates the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- SB.SBÜ. Van Eğitim ve Araştırma Hastanesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not plan to share your IPD with other researchers.